CLINICAL TRIAL: NCT00292123
Title: Combined Behavioral and Pharmacologic Treatment of Polydrug Abuse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Kenzie L. Preston, Ph.D., Principal Investigator, National Institute on Drug Abuse
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDAIRP 326
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-12

CONDITIONS: Opioid Dependence; Cocaine Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Cocaine-Related Disorders | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methadone
Behavioral: Contingency Management

SUMMARY:
The primary goal of this study is to determine how contingency management can best be combined with standard or high doses of methadone to increase simultaneous abstinence from heroin and cocaine.

DETAILED DESCRIPTION:
A study of people pmaintained on Methadone using contingency management

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependence; cocaine use

Exclusion Criteria:

* Medical or psychiatric conditions that would contraindicate participation in a methadone maintenance study; inability to give informed consent; inability to attend clinic seven days a week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 1999-06; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, PhD, Principal Investigator — NIFA Intramural Research Program

REFERENCES:
- [Result] Ghitza UE, Epstein DH, Preston KL. Contingency management reduces injection-related HIV risk behaviors in heroin and cocaine using outpatients. Addict Behav. 2008 Apr;33(4):593-604. doi: 10.1016/j.addbeh.2007.11.009. Epub 2007 Nov 17. PMID 18068905
- [Result] Willner-Reid J, Belendiuk KA, Epstein DH, Schmittner J, Preston KL. Hepatitis C and human immunodeficiency virus risk behaviors in polydrug users on methadone maintenance. J Subst Abuse Treat. 2008 Jul;35(1):78-86. doi: 10.1016/j.jsat.2007.08.011. Epub 2007 Oct 10. PMID 17931826
- [Result] Ghitza UE, Epstein DH, Schmittner J, Vahabzadeh M, Lin JL, Preston KL. Randomized trial of prize-based reinforcement density for simultaneous abstinence from cocaine and heroin. J Consult Clin Psychol. 2007 Oct;75(5):765-74. doi: 10.1037/0022-006X.75.5.765. PMID 17907858
- [Result] Ghitza UE, Epstein DH, Preston KL. Psychosocial functioning and cocaine use during treatment: strength of relationship depends on type of urine-testing method. Drug Alcohol Depend. 2007 Dec 1;91(2-3):169-77. doi: 10.1016/j.drugalcdep.2007.05.018. Epub 2007 Jul 10. PMID 17624688
- [Result] Heinz A, Epstein DH, Preston KL. Spiritual/Religious experiences and in-treatment outcome in an inner-city program for heroin and cocaine dependence. J Psychoactive Drugs. 2007 Mar;39(1):41-9. doi: 10.1080/02791072.2007.10399863. PMID 17523584
- [Result] Heinz AJ, Epstein DH, Schroeder JR, Singleton EG, Heishman SJ, Preston KL. Heroin and cocaine craving and use during treatment: measurement validation and potential relationships. J Subst Abuse Treat. 2006 Dec;31(4):355-64. doi: 10.1016/j.jsat.2006.05.009. Epub 2006 Aug 1. PMID 17084789
- [Result] Ghitza UE, Epstein DH, Preston KL. Nonreporting of cannabis use: Predictors and relationship to treatment outcome in methadone maintained patients. Addict Behav. 2007 May;32(5):938-49. doi: 10.1016/j.addbeh.2006.06.034. Epub 2006 Aug 1. PMID 16887281